CLINICAL TRIAL: NCT01407796
Title: PET Imaging of Endotoxin-induced iNOS Activation in Healthy Volunteers
Brief Title: PET Imaging of Endotoxin-induced iNOS Activation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other)
Responsible Party: Principal Investigator, Delphine L. Chen, MD, Assistant Professor of Radiology, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BJHF/ICTS 7326-01
Record Dates: First submitted 2011-07-28; First posted 2011-08-02 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Pneumonia
Keywords: lung inflammation; positron emission tomography (PET); fluorodeoxyglucose (FDG); inducible nitric oxide synthase (iNOS); lung anti-inflammatory therapy
MeSH Terms: conditions — Pneumonia | interventions — Endotoxins; Lipopolysaccharides; Fluorine-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endotoxin and [18F](+/-)NOS (Experimental): All volunteers in this study will receive endotoxin in a single segment of the lung to induce mild, self-limited inflammation. They will also be imaged before and after endotoxin instillation with the novel PET tracer F-18 (+/-) NOS
  Interventions: Drug: Endotoxin (E. coli O:113, Reference Endotoxin); Drug: [18F](+/-)NOS

INTERVENTIONS:
Drug: Endotoxin (E. coli O:113, Reference Endotoxin)
  Other Names: Lipopolysaccharide
Drug: [18F](+/-)NOS

SUMMARY:
The overall purpose of this research is to gain understanding of the basic responses of the lung to inflammation. Inflammation is the way our bodies react to irritation or injury, and involves red, warm, and often painful swelling of the affected tissue. "Acute lung injury" involves a generalized inflammation to the lung that is activated by any of several conditions: infection, trauma, inhalation of toxic substances, etc. When lung injury is severe, not enough oxygen can get into the body; this can lead to the need for mechanical support of breathing (mechanical ventilation), problems with brain, heart or other organ function, and in some cases, death. Inducible nitric oxide synthase (iNOS) contributes to the development of lung inflammation.

DETAILED DESCRIPTION:
The investigators plan to use [18F](+/-)NOS (the F stands for fluorine and NOS stands for Nitric Oxide Synthase, the name for the investigational radioactive drug that targets iNOS) and positron emission tomography (PET) imaging as a measure of lung inflammation. PET is a machine that detects radiation and generates pictures using a donut shaped scanner similar in appearance to an x-ray "CAT" scan.

In order to show that [18F](+/-)NOS-PET is related to the amount of inflammation, the investigators first need to create a state of controlled lung inflammation that can be measured and quantified. "Controlled lung inflammation" means a reaction in the lungs that is similar to that which occurs during lung infection (increased respiratory secretions, and cough). It is "controlled" because the investigators will not be using anything alive or contagious (it will not spread from one part of your body to another, and cannot spread to another person) and a small area in only one lung will be affected. In order to create this state of controlled lung inflammation, the investigators plan to put a small amount of endotoxin into a single small section of the lung using a bronchoscope (a long, flexible, narrow tube that is passed through the nose or the mouth into the airways of the lung). This use of endotoxin is considered investigational. The investigators have received permission from the FDA to use endotoxin in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man or woman, any race or ethnicity, age 19 - 44 years old
* Screening Pulmonary Function Test
* Screening oxygen saturation by pulse oximetry >97% on room air
* Capable of lying still and supine within the PET/CT scanner for 1.5 hours
* Capable of following instructions for breathing protocol during CT portion of PET/CT
* Able and willing to give informed consent
* BMI < 35

Exclusion Criteria:

* Pregnancy (confirmed by qualitative serum hCG pregnancy test)
* Lactation
* Active menstruation
* History of cardiopulmonary disease
* Currently taking any prescription medications
* History of tobacco use or illicit drug use within the past year
* Presence of implanted electronic medical device
* Enrollment in another research study of an investigational drug
* Known allergy to both trimethoprim/sulfamethoxazole and amoxicillin
* Known allergy to drugs routinely used during bronchoscopy
* Inability lie flat for 1.5 hours for PET/CT scans or follow breathing protocol instructions for the CT portion of the PET/CT

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Distribution volume ratio (DVR), determined by Logan plot analysis, in the right middle lobe. | Change in DVR on post-endotoxin scan (Day 2) from baseline (Day 1).

SECONDARY OUTCOMES:
Bronchoalveolar lavage (BAL) fluid cell counts. | 24 hours after endotoxin instillation.
  Total nucleated and neutrophil cell counts obtained by BAL after endotoxin instillation.
Number and percent of iNOS-stained BAL cells. | 24 hours after endotoxin instillation.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine L. Chen, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicne, St Louis, Missouri, United States

REFERENCES:
- [Derived] Huang HJ, Isakow W, Byers DE, Engle JT, Griffin EA, Kemp D, Brody SL, Gropler RJ, Miller JP, Chu W, Zhou D, Pierce RA, Castro M, Mach RH, Chen DL. Imaging pulmonary inducible nitric oxide synthase expression with PET. J Nucl Med. 2015 Jan;56(1):76-81. doi: 10.2967/jnumed.114.146381. Epub 2014 Dec 18. PMID 25525182